CLINICAL TRIAL: NCT00628732
Title: A Pharmacokinetic and Phase II Study of Oral Cyclophosphamide and Oral Topotecan in Children With Recurrent and or Refractory Solid Tumors
Brief Title: A Pharmacokinetic Study of Oral Cyclophosphamide and Topotecan in Children With Recurrent Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Medical Center Dallas (Other)
Collaborators: Metabolic Solutions Inc. (Industry); Simmons Cancer Center (Other)
Responsible Party: Daniel C. Bowers M.D./ Associate Professor of Pediatrics, UT Southwestern Medical Center of Dallas
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 012005004
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Solid Tumors
Keywords: Cyclophosphamide; Topotecan; Phase II; Children; Relapsed solid tumors
MeSH Terms: interventions — Cyclophosphamide; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Cyclophosphamide and Topotecan

INTERVENTIONS:
Drug: Cyclophosphamide and Topotecan — Two courses of cyclophosphamide at 50 mg/m2/dose and topotecan 0.8 mg/m2/dose by mouth every morning for 14 days each.
  Other Names: Cytoxan and Hycamptin

SUMMARY:
The purposes of this study include:

* Determination of the change in clearance of topotecan and topotecan lactone between day 1 and day 14 for patients receiving treatment with p.o. topotecan and p.o. cyclophosphamide x 14 days.
* Determination of the correlation between the activity of CYP3A4, as measured by the 14C- Erythromycin Breath Test (ERMBT), and topotecan/topotecan lactone clearance for patients receiving treatment with p.o. topotecan and p.o. cyclophosphamide x 14 days.
* Determination of the response rate to oral cyclophosphamide and oral topotecan in recurrent and/or refractory pediatric solid tumors.
* Obtain additional safety data for the chemotherapy regimen, p.o. topotecan and p.o. cyclophosphamide x 14 days.
* Report the frequency of severe toxicities associated with the level of CYP3A4 activity, as measured by the ERMBT, for patients receiving treatment with p.o. topotecan and p.o. cyclophosphamide x 14 days.

DETAILED DESCRIPTION:
Upon obtaining informed consent, patients will begin two courses of oral cyclophosphamide and topotecan x 14 days. During the first of two courses, patients will perform the 14C-Erythromycin Breath Test and have topotecan pharmacokinetics performed on day 1 and 14. The subjects will also have various medical tests and procedures performed that are part of regular cancer care which include: Medical history and physical examination to be done weekly, blood tests to be done weekly, heart and kidney function tests, various scans to be done after two courses of treatment, and a pregnancy test for females of childbearing age to be done prior to starting treatment.

Patients may continue to receive additional courses of oral cyclophosphamide and topotecan provided that they do not experience tumor progression or intolerable side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be less than 22 years of age inclusive
2. Tumor histologies: medulloblastoma/PNET, neuroblastoma, sarcomas, and other pediatric solid tumors for which there is no known effective therapy.
3. Patients must have measurable disease, documented by clinical, radiographic, or histologic criteria.
4. Patients must have a performance status of 0, 1 or 2. Use Karnofsky for patients > 16 years of age and Lansky for patients <= 16 years of age.
5. Patients must have a life expectancy of >= 8 weeks.
6. Prior Therapy: Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.
7. Patients must not be taking the following medications: growth factors, steroids, and CYP3A4 inducers or inhibitors.
8. Patients must have adequate bone marrow, renal, liver function, pulmonary, or central nervous system function.
9. Must be able and willing to participate in all study procedures, including the ERMBT and pharmacokinetic studies.
10. All patients and/or their parents or legal guardians must sign a written informed consent. (11) All institutional, FDA, and NCI requirements for human studies must be met.

Exclusion Criteria:

1. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
2. Patients with an uncontrolled infection.
3. Allergy to erythromycin
4. Patients who have previously received either cyclophosphamide or topotecan are eligible for this study.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2005-01; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Radiographic imaging | Every 2 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C Bowers, MD, Principal Investigator — UT Southwestern Medical Center of Dallas
Locations (1):
- Children's Medical Center Dallas, Dallas, Texas, United States